CLINICAL TRIAL: NCT01169675
Title: BIBW 2992 Phase I Combination With Pemetrexed in Advanced Solid Tumours
Brief Title: BIBW 2992 (Afatinib) in Combination With Pemetrexed in Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.92
Record Dates: First submitted 2010-07-19; First posted 2010-07-26 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib; Pemetrexed

ARMS (6):
- BIBW 2992 low dose (Experimental): patient receives low dose tablet BIBW 2992 po daily plus pemetrexed 500mg/m^2 on day 1 of 21 day cycle
  Interventions: Drug: BIBW 2992 low dose; Drug: pemetrexed
- BIBW 2992 medium dose (Experimental): patient receives medium dose BIBW 2992 po daily plus pemetrexed 500mg/m^2 on day 1 of 21 day cycle
  Interventions: Drug: pemetrexed; Drug: BIBW 2992 medium dose
- BIBW 2992 high dose (Experimental): patient receives high dose BIBW 2992 po daily plus pemetrexed 500mg/m^2 on day 1 of 21 day cycle
  Interventions: Drug: BIBW 2992 high dose; Drug: pemetrexed
- BIBW 2992 low dose 6 day (Experimental): patient receives low dose BIBW 2992 po daily on days 1-6 plus pemetrexed 500mg/m^2 on day 1 of 21 day cycle
  Interventions: Drug: pemetrexed; Drug: BIBW 2992 low dose 6 day
- BIBW 2992 medium dose 6 day (Experimental): patient receives medium BIBW 2992 po daily on days 1-6 plus pemetrexed 500mg/m^2 on day 1 of 21 day cycle
  Interventions: Drug: pemetrexed; Drug: BIBW 2992 medium dose 6 day
- BIBW 2992 high dose 6 day (Experimental): patient receives high dose BIBW 2992 po daily on days 1-6 plus pemetrexed 500mg/m^2 on day 1 of 21 day cycle
  Interventions: Drug: BIBW 2992 high dose 6 day; Drug: pemetrexed

INTERVENTIONS:
Drug: BIBW 2992 low dose — patient receives low dose BIBW 2992 po daily on day 1 of 21 day cycle
  Arms: BIBW 2992 low dose
Drug: BIBW 2992 high dose — patient receives high dose BIBW 2992 po daily on day 1 of 21 day cycle
  Arms: BIBW 2992 high dose
Drug: pemetrexed — given intravenously on day 1 of a 21 day cycle
  Arms: BIBW 2992 medium dose
Drug: pemetrexed — given intravenously on day 1 of a 21 day cycle
  Arms: BIBW 2992 low dose
Drug: BIBW 2992 high dose 6 day — patient receives high dose BIBW 2992 po daily on days 1-6 on 1 of 21 day cycle
  Arms: BIBW 2992 high dose 6 day
Drug: pemetrexed — given intravenously on day 1 of a 21 day cycle
  Arms: BIBW 2992 low dose 6 day
Drug: pemetrexed — given intravenously on day 1 of a 21 day cycle
  Arms: BIBW 2992 high dose 6 day
Drug: pemetrexed — given intravenously on day 1 of a 21 day cycle
  Arms: BIBW 2992 medium dose 6 day
Drug: pemetrexed — given intravenously on day 1 of a 21 day cycle
  Arms: BIBW 2992 high dose
Drug: BIBW 2992 low dose 6 day — patient receives low dose BIBW 2992 po daily on days 1-6 on day 1 of 21 day cycle
  Arms: BIBW 2992 low dose 6 day
Drug: BIBW 2992 medium dose 6 day — patient receives medium dose BIBW 2992 po daily on day1 to 6 of a 21 day cycle
  Arms: BIBW 2992 medium dose 6 day
Drug: BIBW 2992 medium dose — patient receives medium dose BIBW 2992 po daily on day 1 of 21 day cycle
  Arms: BIBW 2992 medium dose

SUMMARY:
This Phase I study will investigate the safety of BIBW 2992 in combination with standard dose pemetrexed (500mg/m2) given on a 21 day cycle in patients with advanced solid cancers. BIBW 2992 will be given on two different dose schedules; dosing on days 1-21 and dosing on days 1 to 6 of a 21 day cycle.

The use of epidermal growth factor receptor tyrosine kinase inhibitors (EGFR TKIs), including BIBW 2992 have demonstrated efficacy in solid tumors including non-small cell lung cancer (NSCLC). In addition, pemetrexed has demonstrated efficacy and has been approved as single agent chemotherapy in second-line NSCLC patients with adenocarcinoma. The data obtained from this trial shall allow for a conclusion as to whether BIBW 2992 may be safely administered in advanced cancer patients in combination therapy with pemetrexed.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 or older.
2. Eastern cooperative oncology group performance status of 0-2.
3. Life expectancy of at least 12 weeks.
4. Measurable disease according to Response evaluation criteria in solid tumors 1.1 criteria.
5. Written informed consent

Exclusion criteria:

1. Treatment with an investigational drug within the past 28 days prior to the start of therapy
2. Persisting toxicities which are clinically significant from previous therapy
3. Patients who are unwilling or unable to take folic acid and vitamin B12 supplementation
4. Active brain metastases
5. Other active malignancy diagnosed within the past 3 years
6. Concomitant intercurrent illnesses that would limit compliance with trial requirement
7. Patients unable or unwilling to interrupt concomitant administration of Non-steroidal anti-inflammatory drugs (NSAIDS) as per pemetrexed prescribing information
8. Patients who have received prior therapy with BIBW 2992
9. Left ventricular function by echocardiogram or Multiple gated acquisition scan (MUGA) less than institutional lower limit of normal
10. Absolute neutrophil count (ANC) less than 1,500/mm3
11. Platelet count less than 100,000/mm3
12. Hemoglobin less than 90g/L
13. Total bilirubin less than 26µmol/L
14. Alanine amino transferase (ALT) and/or aspartate amino transferase (AST) greater than 2.5 X ULN, except in case of known liver metastasis where maximum 5 X ULN is acceptable
15. Serum creatinine level greater than 133µmol/L and/or creatinine clearance (measured or calculated) less than 45 ml/min
16. History or recent gastrointestinal bleeding, obstruction or perforation or malabsorption syndrome and must be able to swallow the BIBW 2992 in whole by mouth.
17. History of interstitial lung disease
18. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
19. Pregnancy or breast feeding
20. Known or suspected active alcohol or drug abuse
21. Patients unable to comply with the protocol
22. Has a diagnosis of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
23. Any known hypersensitivity to the trial drugs or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Canada (2):
  - 1200.92.1001 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1200.92.1002 Boehringer Ingelheim Investigational Site, Hamilton, Ontario

REFERENCES:
- [Derived] Chu QS, Sangha R, Hotte SJ, Sergenson G, Schnell D, Chand VK, Hirte HW. A phase I, dose-escalation trial of continuous- and pulsed-dose afatinib combined with pemetrexed in patients with advanced solid tumors. Invest New Drugs. 2014 Dec;32(6):1226-35. doi: 10.1007/s10637-014-0139-9. Epub 2014 Jul 19. PMID 25037863

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Afatinib 30 mg: Continuous Afatinib 30 mg plus Pemetrexed. Afatinib is the same intervention as BIBW 2992.
- Continuous Afatinib 40 mg: Continuous Afatinib 40 mg plus Pemetrexed. Afatinib is the same intervention as BIBW 2992.
- Pulsed Afatinib 50 mg: Pulsed Afatinib 50 mg plus Pemetrexed. Afatinib is the same intervention as BIBW 2992.
- Pulsed Afatinib 60 mg: Pulsed Afatinib 60 mg plus Pemetrexed. Afatinib is the same intervention as BIBW 2992.
- Pulsed Afatinib 70 mg: Pulsed Afatinib 70 mg plus Pemetrexed. Afatinib is the same intervention as BIBW 2992.
Period: Overall Study
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg
Started | 20 | 3 | 7 | 17 | 6
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 20 | 3 | 7 | 17 | 6
Not completed — Progressive disease | 13 | 2 | 5 | 15 | 1
Not completed — Dose Limiting Toxicity (DLT) | 1 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 5 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 2
Not completed — Other Reason Not Defined Above | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set includes all randomized patients that received Afatinib or Pemetrexed
Groups:
- Continuous Afatinib 30 mg: Continuous Afatinib 30 mg plus Pemetrexed
- Continuous Afatinib 40 mg: Continuous Afatinib 40 mg plus Pemetrexed
- Pulsed Afatinib 50 mg: Pulsed Afatinib 50 mg plus Pemetrexed
- Pulsed Afatinib 60 mg: Pulsed Afatinib 60 mg plus Pemetrexed
- Pulsed Afatinib 70 mg: Pulsed Afatinib 70 mg plus Pemetrexed
- Total: Total of all reporting groups
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg | Total
Number analyzed (Participants) | 20 | 3 | 7 | 17 | 6 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.4) | 53.7 (16.6) | 69.6 (10.5) | 57.9 (10.7) | 64.8 (7.4) | 60.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 1 | 11 | 2 | 27
  Male | 9 | 1 | 6 | 6 | 4 | 26

OUTCOME MEASURES:

1. Primary Outcome: Investigator Defined Dose Limiting Toxicity (DLT) During First Course of Treatment, Treated Set
Description: Occurence of DLT during the first course of treatment to determine the maximum tolerated dose (MTD) of Afatinib at two different dose schedules in combination with the standard established dose of pemetrexed (500 mg/m2).
Time Frame: DLT were assessed during the first cycle (days 1-21)
Population: Treated Set includes all patients that received treatment of Afatinib or Pemetrexed that who were evaluable for MTD determination
Measure: Number; unit: participants
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg
Number analyzed (Participants) | 19 | 3 | 6 | 17 | 6
participants | 6 | 2 | 1 | 6 | 4

2. Secondary Outcome: Investigator Defined Dose Limiting Toxicity (DLT) During All Courses of Treatment, Treated Set
Description: Occurence of DLT during all courses of treatment with Afatinib at two different dose schedules in combination with the standard established dose of pemetrexed (500 mg/m2).
Time Frame: DLT were assessed during all cycles of treatment
Population: Treated Set includes all patients that received treatment of Afatinib or Pemetrexed
Measure: Number; unit: participants
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg
Number analyzed (Participants) | 20 | 3 | 7 | 17 | 6
participants | 11 | 2 | 3 | 11 | 4

3. Secondary Outcome: Objective Response (OR)
Description: Objective Response is defined as complete response or partial response according to the response evaluation criteria in solid tumours (RECIST) version 1.1.
  Complete Response (CR): disappearance of all non-target lesions and normalization of tumor marker level; Partial Response (PR): at least 30% decrease of the sum of longest diameter (LD) of target lesions; Progressive Disease (PD): at least a 20% increase in the sum of LD of target lesions together with an absolute increase in the sum of LD of at least 5 millimeters; Stable Disease (SD): neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD.
Time Frame: Every 6 weeks before week 48 and every 12 weeks after week 48 until progression
Population: Treated Set includes all patients that received treatment of Afatinib or Pemetrexed
Measure: Number; unit: participants
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg
Number analyzed (Participants) | 20 | 3 | 7 | 17 | 6
participants | 2 | 0 | 0 | 2 | 0

4. Secondary Outcome: Disease Control
Description: Disease Control is defined as complete response, partial response, or stable disease according to the response evaluation criteria in solid tumours (RECIST) version 1.1.
Time Frame: Every 6 weeks before week 48 and every 12 weeks after week 48 until progression
Population: Treated Set includes all patients that received treatment of Afatinib or Pemetrexed
Measure: Number; unit: participants
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg
Number analyzed (Participants) | 20 | 3 | 7 | 17 | 6
participants | 6 | 1 | 3 | 6 | 2

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first treatment to the occurence of tumour progression or death, whichever came first. It was assessed according to RECIST version 1.1 criteria.
Time Frame: Every 6 weeks before week 48 and every 12 weeks after week 48 until progression
Population: Treated Set includes all patients that received treatment of Afatinib or Pemetrexed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg
Number analyzed (Participants) | 20 | 3 | 7 | 17 | 6
months | 2.49 [1.21 to 3.97] | 2.52 [1.14 to 5.32] | 2.56 [1.21 to 6.50] | 2.52 [1.21 to 4.13] | 2.69 [0.82 to 7.85]

6. Secondary Outcome: Tumour Shrinkage
Description: Tumour shrinkage is defined as the maximum percentage decrease from baseline in the sum of the longest diameters of target lesions.
Time Frame: Every 6 weeks before week 48 and every 12 weeks after week 48 until progression
Population: Treated Set: all patients that received treatment of Afatinib or Pemetrexed and who were evaluated for the longest diameter of the target lesions.
Measure: Number; unit: participants
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg
Number analyzed (Participants) | 17 | 2 | 7 | 16 | 3
participants
  Patients with any decrease in tumour size | 10 | 2 | 3 | 5 | 1
  Patients having >30% decrease in tumour size | 2 | 0 | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Starting with first administration of trial drug (Afatinib or Pemetrexed) and ending 28 days after the last administration of trial drug.
Arm/Group | Continuous Afatinib 30 mg | Continuous Afatinib 40 mg | Pulsed Afatinib 50 mg | Pulsed Afatinib 60 mg | Pulsed Afatinib 70 mg
Serious Adverse Events (participants affected / at risk) | 9/20 | 2/3 | 3/7 | 4/17 | 4/6
Other Adverse Events (participants affected / at risk) | 20/20 | 3/3 | 7/7 | 17/17 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Afatinib 30 mg (N=20) | Continuous Afatinib 40 mg (N=3) | Pulsed Afatinib 50 mg (N=7) | Pulsed Afatinib 60 mg (N=17) | Pulsed Afatinib 70 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Intestinal prolapse (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous Afatinib 30 mg (N=20) | Continuous Afatinib 40 mg (N=3) | Pulsed Afatinib 50 mg (N=7) | Pulsed Afatinib 60 mg (N=17) | Pulsed Afatinib 70 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 10 | 1 | 5 | 10 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 1 | 1 | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 3 | 1 | 1 | 0 | 0
Eye discharge (Eye disorders) | 2 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 2 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 0 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 2 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Aptyalism (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 7 | 0 | 5 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 3 | 5 | 14 | 6
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 0 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Intestinal prolapse (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 2 | 4 | 13 | 5
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 15 | 3 | 6 | 11 | 5
Vomiting (Gastrointestinal disorders) | 9 | 1 | 5 | 11 | 3
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 1 | 0
Chills (General disorders) | 3 | 1 | 1 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 18 | 2 | 7 | 16 | 5
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 3 | 4 | 2
Pain (General disorders) | 3 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 5 | 0 | 4 | 3 | 3
Thirst (General disorders) | 0 | 1 | 1 | 0 | 0
Unevaluable event (General disorders) | 0 | 0 | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 4 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 2 | 0
Omphalitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 1 | 1 | 3 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 0 | 6 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 1 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 5 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 2 | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 | 0 | 1 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 9 | 1 | 4 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 16 | 3 | 5 | 13 | 6
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 2 | 3 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0 | 1 | 7 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3 | 5 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 3 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 2 | 3 | 2
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 2 | 2
Headache (Nervous system disorders) | 3 | 0 | 1 | 3 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 1 | 1 | 3 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 0 | 1 | 3 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 0 | 1 | 3 | 3
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 3 | 1 | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Penile discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 2 | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 4 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 1 | 3 | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 0 | 0
Hangnail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 2 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 0 | 3 | 4 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 4 | 3 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 13 | 3 | 5 | 15 | 5
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 3 | 1 | 0 | 3 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.